CLINICAL TRIAL: NCT06647966
Title: Diagnostic Performance of [11C]Choline PET/CT In the Preoperative Assessment of Primary Hyperparathyroidism
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiti Arturo, Professor in Diagnostic Imaging and Radiotherapy Faculty of Medicine and Surgery, Vita-Salute San Raffaele University Director, Department of Nuclear Medicine, IRCCS Ospedale San Raffaele, IRCCS San Raffaele
Other Study IDs: CHOPET-HYPER
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Primary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Primary | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with clinical signs of hyperparathyroidism
  Interventions: Diagnostic Test: PET/CT

INTERVENTIONS:
Diagnostic Test: PET/CT — [11C]CH PET/CT

SUMMARY:
Primary hyperparathyroidism (HPT) ranks as the third most common endocrine disorder, characterized by excessive secretion of parathormone (PTH), a hormone crucial for regulating calcium and phosphorus metabolism within the body. The only cure for HPT is surgically removing the hyperfunctioning parathyroid tissue, both in symptomatic and asymptomatic settings. With the advance of preoperative medical imaging techniques, a paradigm shift has taken place in the surgical approach of this condition, evolving from an inpatient bilateral cervical exploration to an outpatient minimally invasive procedure, which has proved to be superior in outcome. Due to the small size of the glands, preoperative visualisation and localisation are mandatory for the surgeon. Several imaging methods have been researched for identifying hyperfunctioning parathyroid glands, including morphological, functional and hybrid techniques, with no clear agreement on the optimal imaging approach.The preoperative localization modalities available are ultrasonography; parathyroid scintigraphy using technetium [99mTc]Tc sestamibi (MIBI), multiphase multidetector 4D computed tomography (4DCT); magnetic resonance imaging; and recently, positron-emission tomography/computed tomography (PET/CT) using 11C- and 18F-labelled radiotracers. While ultrasound and [99mTc]Tc-MIBI scintigraphy have been long used to diagnose and monitor patients with HPT, they can lead to numerous false negative results and therefore require additional examinations.Choline PET/CT is steadily replacing conventional imaging in many centres, allowing for the localization of adenomas in three quarter of patients with negative previous imaging examinations, but is still considered a relatively new method. [11C]C-Choline ([11C]CH) PET/CT is gradually gaining ground as a reliable method of localising HPT preoperatively, due to its fast uptake in hyperfunctioning parathyroid tissue, shorter acquisition time and lower radiation exposure compared to other nuclear medicine investigations and conventional methods. [11C]CH PET/CT has been suggested to be superior in diagnostic performances, compared to other imaging methods, reaching sensitivities up to 98.9%.The aim of our retrospective, single centre study is to evaluate the diagnostic performances and the inter-observer agreement of [11C]CH PET/CT for the preoperative detection of parathyroid adenomas in patients with suspected primary HPT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biochemically proven HPT, either through elevated serum levels of PTH or normal PTH despite hypercalcemia;
* Age ≥ 18 years old;
* [11C]CH PET/CT for HPT before eventual surgery.

Exclusion Criteria:

* Pregnancy or breast-feeding.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Retrospectively select patients who performed PET in our institution from 2022 until 2024.
  Patients who meet the following criteria will be included in the study.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the diagnostic performances of [11C]CH PET/CT in patients with biochemically proven HPT. | [11C]CH PET/CT : day 0
  Calculation of diagnostic performance parameters: sensitivity, specificity, accuracy, positive and negative predictive values.

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Chiti, MD, Study Director — IRCCS Ospedale San Raffaele
Locations (1):
- Irccs San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No